CLINICAL TRIAL: NCT02419573
Title: Pragmatic Trial of Airway Management in Out-of-Hospital Cardiac Arrest
Brief Title: Pragmatic Airway Resuscitation Trial
Acronym: PART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Henry E. Wang, MD, MS, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL077863-PART; 5U01HL077863 (NIH); UH2HL125163 (NIH)
Record Dates: First submitted 2015-02-25; First posted 2015-04-17 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation; laryngeal tube; endotracheal intubation; non-traumatic Out of Hospital Cardiac Arrest (OOHCA)
MeSH Terms: conditions — Heart Arrest | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotracheal Intubation (Active Comparator): The insertion of a plastic breathing tube through the mouth and into the trachea.
  Interventions: Device: Endotracheal Intubation
- Laryngeal Tube (King) (Active Comparator): Insertion of a supraglottic airway (SGA)
  Interventions: Device: Laryngeal Tube (King)

INTERVENTIONS:
Device: Endotracheal Intubation — In this traditional model of OHCA airway management, advanced-level Emergency Medical Services (EMS) personnel will use ETI as the primary (initial) airway management intervention. If the EMS agency is assigned to this arm, basic-level EMS personnel will use bag-valve-mask ventilation only even if they would normally use an LT.
  Arms: Endotracheal Intubation
Device: Laryngeal Tube (King) — In this test model of OHCA airway management, advanced-level Emergency Medical Services (EMS) personnel will use LT as the primary (initial) airway management intervention. Basic-level EMS personnel will use bag-valve-mask ventilation. If trained to use LT, basic-level EMS personnel may perform LT insertion.
  Other Names: King (LT-D); King (LTS-D); King (LT)
  Arms: Laryngeal Tube (King)

SUMMARY:
The primary objective of the trial is to determine if 72-hour survival after out-of-hospital cardiac arrest (OHCA) is improved with initial endotracheal intubation (ETI) over initial laryngeal tube (LT) airway management strategies.

DETAILED DESCRIPTION:
The primary objective of the trial is to determine if 72-hour survival after out-of-hospital cardiac arrest (OHCA) is improved with initial endotracheal intubation (ETI) over initial laryngeal tube (LT) airway management strategies.

The null hypothesis is that 72-hour survival is similar between primary Laryngeal Tube (LT) SGA and primary ETI airway management strategies.

Evaluated secondary outcomes will include return of spontaneous circulation, survival to hospital discharge, neurologically intact survival at hospital discharge, airway management performance, and clinical adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA)
* Adult (age ≥18 years or per local interpretation)
* Non-traumatic etiology
* Initiation of ventilatory support (e.g., bag-valve-mask device, non-rebreather mas, etc.)

Exclusion Criteria:

* Known pregnant women
* Known prisoners
* Major facial trauma (visible major deformity, copious oral bleeding, etc)
* Major bleeding or exsanguination (e.g., major upper or lower GI bleed, visceral perforation, major uncontrolled bleeding from laceration or injury)
* Patient receiving initial care by a non-PART participating EMS agency capable of performing ETI, LT, or other advanced airway management
* Patients with ET tube, LT or other advanced airway device inserted prior to participating EMS agency arrival (e.g., inserted by healthcare facility personnel)
* Patients with a pre-existing tracheostomy
* Obvious asphyxial cardiac arrest (e.g., choking, foreign body aspiration, angioedema, epiglottitis, trauma to mouth and face, etc.)
* Patients with a left ventricular assist device (LVAD) or total artificial heart (TAH)
* Patients with pre-existing written "do-not-attempt-resuscitation" (DNAR) orders
* Inter-facility transports
* Patients with a "do not enroll" bracelet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3004 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Wang, MD, Principal Investigator — University of Alabama, University of Texas Health Science Center at Houston
Locations (6):
- United States (6):
  - Alabama Resuscitation Center, Birmingham, Alabama
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Cente, Dallas, Texas
  - University of Washington (Data Coordinating Center), Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nassal MMJ, Elola A, Aramendi E, Jaureguibeitia X, Powell JR, Idris A, Raya Krishnamoorthy BP, Daya MR, Aufderheide TP, Carlson JN, Stephens SW, Panchal AR, Wang HE. Temporal Trends in End-Tidal Capnography and Outcomes in Out-of-Hospital Cardiac Arrest: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419274. doi: 10.1001/jamanetworkopen.2024.19274. PMID 38967927
- [Derived] Wang HE, Humbert A, Nichol G, Carlson JN, Daya MR, Radecki RP, Hansen M, Callaway CW, Pedroza C. Bayesian Analysis of the Pragmatic Airway Resuscitation Trial. Ann Emerg Med. 2019 Dec;74(6):809-817. doi: 10.1016/j.annemergmed.2019.05.009. Epub 2019 Jul 2. PMID 31272823
- [Derived] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- See also: Resuscitation Outcomes Consortium (ROC) Public Homepage — http://roc.uwctc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
Started | 1499 | 1505
Completed | 1495 | 1505
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 3,004 enrolled, 3 lost to follow-up, 1 withdrew from study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King) | Total
Number analyzed (Participants) | 1495 | 1505 | 3000
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (16.9) | 63.2 (17.0) | 63.1 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants] — The gender was "unknown" for 1 female patient in LT and 1 male patient in LT.
  Participants
    Female | 598 | 576 | 1174
    Male | 897 | 929 | 1826
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 7 | 10
  Asian | 27 | 35 | 62
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 493 | 385 | 878
  White | 804 | 903 | 1707
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 163 | 170 | 333
Region of Enrollment [Number; unit: participants]
  United States | 1495 | 1505 | 3000

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive at 72 Hours After Episode.
Description: Number of patient alive at 72 hours after episode.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
Number analyzed (Participants) | 1495 | 1505
Participants | 230 | 275

2. Secondary Outcome: Return of Spontaneous Circulation (ROSC)
Description: Presence of palpable pulses on Emergency Department arrival. Patients pronounced dead in the field coded as ROSC=[none].
Time Frame: Patients will be followed from the time of the CA until death or ROSC whichever occurs first. The time frame for this secondary outcome may vary from minutes to hours, but is not expected to last longer than 12 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
Number analyzed (Participants) | 1495 | 1505
Participants | 361 | 420

3. Secondary Outcome: Number of Patients Alive at Hospital Discharge
Description: Number of patients alive at time hospital discharge.
Time Frame: From enrollment through end of hospital course. Maximum time interval not specified. Maximum time interval observed in study was 138 days.
Population: Outcome for 1 patient in LT group not known.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
Number analyzed (Participants) | 1495 | 1504
Participants | 121 | 163

4. Secondary Outcome: Number of Patients With Favorable Neurologic Status on Hospital Discharge
Description: Number of patients with favorable neurologic status, defined as Modified Rankin Scale (MRS) <=3.
  MRS values for neurologic outcome include:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: From enrollment through end of hospital course.
Population: Neurologic status not known for 4 patients in the ETI group and 5 patients in LT group.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
Number analyzed (Participants) | 1495 | 1500
Participants | 75 | 107

ADVERSE EVENTS:
Time Frame: 72 hours of hospitalization.
Arm/Group | Endotracheal Intubation | Laryngeal Tube (King)
All-Cause Mortality (participants affected / at risk) | 1265/1495 | 1230/1505
Serious Adverse Events (participants affected / at risk) | 0/1495 | 0/1505
Other Adverse Events (participants affected / at risk) | 582/1495 | 173/1505
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Endotracheal Intubation (N=1495) | Laryngeal Tube (King) (N=1505)
Multiple (>=3) attempts to insert the assigned airway. (Injury, poisoning and procedural complications) | 245/1299 (245) | 61/1353 (61) — Multiple attempts (>=3) to insert the assigned airway device. Based upon EMS personnel report.
Unsuccessful insertion of assigned airway. (Injury, poisoning and procedural complications) | 573/1299 (573) | 159/1353 (159) — Unsuccessful efforts to insert the assigned airway device. Based upon EMS personnel reports.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 30/426 (30) | 17/485 (17) — Pneumothorax detected on first chest x-ray. Based upon radiology reports.
Rib Fracture (Respiratory, thoracic and mediastinal disorders) | 30/426 (30) | 16/85 (16) — Rib fractures detected on first chest x-ray. Based upon Radiology reports.
Pneumonia or Aspiration Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 89/398 (89) | 120/460 (120) — Pneumonia or aspiration pneumonitis reported during first 72 hours of hospitalization. Based upon radiology reports.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT02419573/Prot_SAP_000.pdf